CLINICAL TRIAL: NCT05789394
Title: Phase 1, Dose Escalation, Non-Randomized, Open Label, Clinical Trial Evaluating the Safety and Preliminary Efficacy of Allogenic Adipose-Derived Mesenchymal Stem Cells (AMSCs) for Recurrent Glioblastoma
Brief Title: Allogenic Adipose-Derived Mesenchymal Stem Cells for the Treatment of Recurrent Glioblastoma or Recurrent Astrocytoma in Patients Undergoing Craniotomy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC220704; NCI-2023-02057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-004561 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Glioblastoma, IDH-Wildtype; Recurrent Astrocytoma, IDH-Mutant, Grade 4; Astrocytoma, Grade IV
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Specimen Handling; Craniotomy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AMSCs) (Experimental): Patients receive AMSCs IT and undergo Ommaya reservoir placement during a craniotomy on study. Patients also undergo MRI on study and during follow-up, as well as blood sample, tissue sample, and CSF sample collection on study.
  Interventions: Biological: Allogeneic Adipose-derived Mesenchymal Stem Cells; Procedure: Biospecimen Collection; Procedure: Craniotomy; Procedure: Magnetic Resonance Imaging; Procedure: Ommaya Reservoir Tap

INTERVENTIONS:
Biological: Allogeneic Adipose-derived Mesenchymal Stem Cells — Receive IT
  Other Names: Allogeneic Adipose-derived MSCs; Allogeneic Adipose-derived Stem/Stromal Cells; Allogeneic Mesenchymal Stem/Stromal Cells
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Craniotomy — Undergo craniotomy
  Other Names: incision of the skull; Open Craniotomy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); MRIs; sMRI; Structural MRI
Procedure: Ommaya Reservoir Tap — Undergo Ommaya reservoir placement for collection of CSF
  Other Names: Ommaya Reservoir Access

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of allogenic adipose-derived mesenchymal stem cells (AMSCs) in treating patients with glioblastoma or astrocytoma that has come back (recurrent) who are undergoing brain surgery (craniotomy). Glioblastoma is the most common and most aggressive form of primary and malignant tumor of the brain. Currently, the standard of care for this disease includes surgical resection, followed by radiation with chemotherapy and tumor treating fields. Despite this aggressive therapy, the survival after finishing treatment remains low and the disease often reoccurs. Unfortunately, the available therapy options for recurrent glioblastoma are minimal and do not have a great effect on survival. AMSCs are found in body fat and when separated from the fat, are delivered into the surgical cavity at the time of surgery. When in direct contact with tumor cells, AMSCs affect tumor growth, residual tumor cell death, and chemotherapy resistance. The use of AMSCs delivered locally into the surgical cavity of recurrent glioblastoma during a craniotomy could improve the long-term outcomes of these patients by decreasing the progression rate and invasiveness of malignant cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the maximum tolerated dose (MTD) of locally delivered adipose-derived mesenchymal stem cells (AMSCs) in patients with recurrent glioblastoma (GBM).

SECONDARY OBJECTIVES:

I. To assess the safety and toxicity profile of locally delivered AMSCs in patients with recurrent GBM.

II. To assess overall survival (OS) in recurrent GBM patients treated with locally delivered AMSCs.

III. To assess progression free survival (PFS) in recurrent GBM patients treated with locally delivered AMSCs.

CORRELATIVE OBJECTIVES:

I. To explore the systemic immune response after application of AMSCs through cytokine analysis on peripheral blood samples.

II. To explore the local changes on the brain parenchyma by analyzing tissue at recurrence.

III. To explore the presence of AMSCs on brain tissue at recurrence.

OUTLINE: This is a dose-escalation study.

Patients receive AMSCs intratumorally (IT) and undergo Ommaya reservoir placement during a craniotomy on study. Patients also undergo magnetic resonance imaging (MRI) on study and during follow-up, as well as blood sample, tissue sample and cerebrospinal fluid (CSF) sample collection on study.

After completion of study treatment patients are followed up every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants >= 18 years
* Karnofsky Performance Scale (KPS) >= 60
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Patients with a previous histological diagnosis of glioblastoma multiforme, isocitrate dehydrogenase (IDH) wildtype (WT) or astrocytoma, IDH-mutant World Health Organization (WHO) grade IV according to the 2021 WHO classification of tumors of the central nervous system , who are candidates to- and will undergo a redo craniotomy for excision of recurrent tumor
* There is measurable disease according to the immunotherapy response assessment in neuro-oncology (iRANO) criteria
* Serum creatinine and urea <= 2 times the upper limit of normal (=< 3 weeks prior to registration)
* Alanine transaminase (ALT), aspartate transferase (AST) and alkaline phosphatase =< 3 times the upper limit of normal, and bilirubin =< 2.5 mg/dL (=< 3 weeks prior to registration)
* Prothrombin time =< 1.5 times upper limit of normal (=< 3 weeks prior to registration)
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 times the upper limit of normal (=< 3 weeks prior to registration)
* Hemoglobin >= 9 g/dL (=< 3 weeks prior to registration)
* Platelets >= 100 x 10^9/L (=< 3 weeks prior to registration)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (=< 3 weeks prior to registration)
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Patient or legally authorized representative (LAR) is able to fully understand and provide written and verbal consent for the protocol
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willingness to undergo Ommaya reservoir placement and provide cerebrospinal fluid (CSF) samples for correlative research

Exclusion Criteria:

* Patients who are undergoing needle biopsy only or non-eligible for a surgical intervention
* Tumors located solely in the brain stem, midbrain, or thalamus without inclusion/involvement of surrounding brain matter
* Previous treatment with bevacizumab
* Radiographic evidence of leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 4 weeks
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients). Will use the standard cohort 3+3 design.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 1 year
  All patients who have received any treatment will be considered evaluable for assessing adverse event rates. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Will follow the Common Terminology Criteria for Adverse Events version 5.0 to record and grade (1-5) any potential AEs.
Best response | Up to 5 years
  Best response per patient is defined to be the best objective status recorded from treatment application until disease progression or death (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Best response assignment will depend on the achievement of both measurement and confirmation criteria.
Response rate (RR) | Up to 5 years
  RR is defined as the number of patients who have achieved complete response or partial response per immunotherapy response assessment for neuro-oncology for recurrent glioblastoma after application of allogeneic adipose-derived mesenchymal stem cells (AMSCs) divided by total number of evaluable patients. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population.
Progression free survival | From time of AMSCs application until the first occurrence of progression or death, assessed up to 5 years
  The quality of survival will be measured by performance status. The data on time-related variables will be summarized descriptively.
Overall survival | From beginning the time of AMSCs application to the date of death, assessed up to 5 years
  The quality of survival will be measured by performance status. The data on time-related variables will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Quinones-Hinojosa, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials